CLINICAL TRIAL: NCT02566148
Title: Life Course, HIV and Hepatitis B Among African Migrants Living in Ile-de-France
Acronym: PARCOURS
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Ministry of Health, France (Other Government); Institut de Recherche pour le Developpement (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut national de prevention et d'education pour la sante (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS PARCOURS
Record Dates: First submitted 2015-06-19; First posted 2015-10-02 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: HIV Infection; Chronic Hepatitis B
Keywords: Life-event survey; observational survey among migrants in France
MeSH Terms: conditions — HIV Infections; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV group: group living with HIV
- Hepatitis B group: group living with chronic hepatitis B
- Reference group: group who has neither HIV nor hepatitis B

SUMMARY:
Populations from Sub-Saharan Africa represent one of the most dynamic immigration flows in France and are among the most exposed to HIV infection and hepatitis B.

The Parcours study aims to understand, among sub-Saharan African migrants, how social and individual factors combine in the course of migration and settlement in France, and influence the risk of infection, access to prevention and care, and the effectiveness of care for both HIV and hepatitis B diseases.

The research was conducted in Ile-de-France, where 60% of sub-Saharan African migrants reside. It consists in a cross-sectional observational survey, using a life-event history approach that reproduces the sequence of different life and health events, and contributes to explain the present situation (type of disease management, patient's quality of life) in light of all the elements of the past trajectory (administrative, familial, socio-economic, professionals).

A representative survey was conducted between February 2012 and May 2013 in health care facilities in Ile-de-France, among three groups of migrants from Sub-Saharan Africa: a group living with HIV, a group living with chronic hepatitis B and a group who has neither of these diseases. For each group, stratified random sampling was used. The survey was conducted in 24 hospital services providing HIV care, 20 health care facilities providing hepatitis B care, and 30 primary health care facilities.

Were eligible all patients attending these health care facilities, born in a Sub-Saharan African country and with Sub-Saharan African citizenship at birth, aged 18 to 59 years, with an HIV diagnosis (HIV group) or chronic hepatitis B diagnosis (hepatitis B group) more than three months prior or not diagnosed with HIV or chronic Hepatitis B (reference group).

Among the patients offered participation, 926 HIV-infected patients, 779 patients infected by hepatitis B, and 763 patients without these two diseases participated in the study.

For all participants, detailed information on socio-demographic characteristics; migration and life conditions in France; social, sexual and reproductive life history; and screening and care history were collected using a life-event history questionnaire administered face-to-face by a specialized interviewer. Health care professionals documented clinical information from the medical records. Data was collected anonymously.

DETAILED DESCRIPTION:
The PARCOURS study was conducted to study how health trajectories and social and migratory paths are interlaced for migrants from sub-Saharan Africa living in France. This retrospective quantitative life-event survey was conducted from February 2012 to May 2013 in health-care facilities in the greater Paris metropolitan area (Ile-de-France), among three groups of migrants born in sub-Saharan Africa: one group receiving HIV care, one group with chronic hepatitis B, and a third group of people visiting primary-care centres. Recruitment took place at facilities randomly selected from an exhaustive list of HIV outpatient hospital clinics (n=24), hepatitis treatment clinics (n=20) and general practice medical centres (n=30).

Recruitment procedure for patients in each group:

Within each health care facility selected for the study, all health care professionals providing outpatient care to patients born in sub-Saharan Africa were asked to participate in the study. They identified eligible patients during consultations based on medical records, and offered study participation to all eligible patients, except when the patient was deemed unable to be interviewed (for mental health or physical health reasons or because were unable to be interviewed in one of the languages spoken by the interviewer). When the patient agreed to participate in the study, health care professionals gave her/him an information leaflet on the study and obtained written consent. They also gave the participant a card bearing an identification number to ensure data collection anonymity and confidentiality, and referred her/him to the Parcours interviewer at the end of the consultation. The Parcours interviewer conducted the interview right after the consultation, in face-to-face mode, in a dedicated room, with closed door to ensure privacy.

The health care professional could also suggest an appointment in the following days, always on site, to patients who agreed to participate in the study but were not immediately available.

Consideration of non-Francophone participants:

To take into account difficulties in participating in the survey due to poor or no knowledge of the French language, the patient questionnaire was available in French or English, and, by appointment, an interpreter could be made available to conduct the interview in an African language spoken by the respondent.

Type of data collected

Several data collection tools were used:

Information register :

In each service investigated, each health care professional participating in the study held an information register. Each page of the register had two parts, one with a detachable section specifying the correspondence between the identity of study patients and their identity number, and an anonymous one describing the main characteristics of eligible patients. During each consultation day, the health care professional listed in the register all eligible patients, their gender, age group, if the patient had worked at least one day in the previous month, a health indicator (last CD4 count for HIV + patients, last alanine transaminase (ALT) level for patients with hepatitis B, the fact of consulting in this facility for the first time for patients in the reference group), and participation in the survey (participant, not offered participation, refusal).

Life-event history questionnaire

Participants were interviewed using a standardized life-event history questionnaire administered by an interviewer face-to-face (average duration 55 minutes). The life-event questionnaire consisted of two parts:

* A list of questions associated with a life event calendar (or biographical grid), which allowed identifying, recording and dating (per year) events in the lives of the respondents, from birth to the date of the survey, and in the various themes explored in the study.
* A book of thematic modules, aimed at describing in-depth the events previously identified in the biographical grid (or some of them).

The life-event calendar has a very graphic and visual form, which makes it easier to remember, record and date the events in the lives of the respondents. In particular, it encourages and easily adapts to the process of remembering that works by association of ideas and connections between life-event areas and as such optimizes data collection, in terms of completeness and reliability of the data collected.

The themes explored in the life-event questionnaire were:

Gender, age ; Residential biography and housing history ; Place of birth and places of residence. ; Work history - Education and Resources ; Marital and family history ; History of testing ; General health and history of disease ; Arrival in France and stay in France ; Sexual and reproductive health ; Social networks, support networks

Medical questionnaire :

The health care professional completed the medical questionnaire, from the patient's medical record. For the HIV and hepatitis B groups, this questionnaire documented the chronological landmarks and key parameters of the disease and its treatment. For the reference group, it informed the reason for consultation, potential diseases at the time of the survey, and current treatments.

Anonymity of data:

The identity number on the anonymity card given by the health care professional to the patient was the only participant identifier for the different survey questionnaires (thematic book and life-event calendar, medical questionnaire). The interviewer did not know the identity of the patient. No personally identifiable data was collected directly or indirectly for eligible individuals not offered participation or individuals refusing study participation. The general characteristics collected on the register among refusals were collected in the form of classes, and not precisely, thus not allowing for later identification.

Ethical approvals :

The survey was approved by the Advisory Committee for Data Processing in Health Research (CCTIRS) (approval on 13 April 2011) and by the National Commission on Informatics and Liberties (CNIL) (CD-2011-484 approval on 7 December 2011).

Data collection :

Between 30/01/2012 and 31/12/2012, 1,829 individuals infected with HIV and meeting the eligibility criteria presented at the participating services, among which 141 were not offered participation by their physician (111 for health reasons and 30 for language problems). Of the 1,688 individuals offered participation, 762 refused or abandoned during the questionnaire. In total, 926 individuals were included.

Between 15/02/2012 and 31/05/2013, 1,169 individuals infected with hepatitis B and meeting the eligibility criteria presented at the participating services, among which 17 were not offered participation by their physician and 8 abandoned during the questionnaire due to language problems. In total, among the 1,135 individuals offered participation, 779 were included.

Between 15/02/2012 and 31/05/2013, 1,184 meeting the eligibility criteria presented at the participating primary health care facilities. Among these, 124 were not offered participation by their physician (91 for health reasons and 33 for language problems). Among the 1,060 individuals offered participation, 297 refused or abandoned during the questionnaire. In total, 763 individuals were included.

Among all services and groups, the number of refusals due to language problems was 71 (30 in HIV group, 8 in Hepatitis B group and 33 in reference group), to which can be added 10 interviews interrupted due to poor understanding of French (8 in hepatitis B group and 2 in reference group).

Weighting :

In order to take into account the sample design and non-participation, data was weighted according to each individual's probability of inclusion in the survey (i.e. considering the probability of inclusion in the sample for each health care facility, the number of half-days of weekly consultations in each facility included and the individual study participation per half-day of included consultations).

ELIGIBILITY:
Inclusion Criteria:

* - For the 3 groups:

  * Be born in a Sub-Saharan African country and with Sub-Saharan African citizenship at birth,
  * Visit the health care facility for one's own health.
* For the HIV group: To have been diagnosed for HIV more than 3 months ago, regardless of co-infections
* For the hepatitis B group: To have been diagnosed with a chronic hepatitis B (AgHBs+) more than 3 months ago and not be HIV co-infected
* For the primary care group: Not be known by the consulting physician as infected by HIV or Hepatitis B.

Exclusion Criteria:

* to have been diagnosed for HIV or hepatitis B less than 3 months ago.
* major cognitive or health impairments

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Migrants from Sub-Saharan Africa living in Ile-de-France (Paris area) and visiting health care facilities: people living with HIV/AIDS (HIV group), people with chronic hepatitis B (hepatitis B group), and people who have neither of these conditions and consult within primary health care facilities in Ile-de-France (reference group).
Sampling Method: Probability Sample
Enrollment: 2468 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Lapse of time from arrival in France to HIV testing | From arrival in France until the date of first HIV testing or date of of data collection, whichever came first, up to 20 years
  Time (in years) to occurence of first HIV testing, from arrival in France
Lapse of time from arrival in France to hepatitis B testing | From arrival in France until the date of first hepatitis B testing or date of of data collection, whichever came first, up to 20 years
  Time (in years) to occurence of first hepatitis B testing, from arrival in France
Lapse of time from HIV diagnostic to access to care | From first HIV diagnostic until the date of entry into care for HIV or date of of data collection, whichever came first, up to 20 years
  Time (in years) to occurence of entry into HIV care, from HIV diagnostic
Lapse of time from hepatitis B diagnostic to access to care | From first hepatitis B diagnostic until the date of entry into care for hepatitis or date of of data collection, whichever came first, up to 20 years
  Time (in years) to occurence of entry into Hepatitis B care, from hepatitis B diagnostic

SECONDARY OUTCOMES:
Condom use | twelve months before data collection
  Systematic condom use during the twelve months before the survey
Evolution in concurrent sexual partnerships after migration in France | At arrival in France, and then each year up to 20 years after arrival in France
  Proportion of the respondents who declared, retrospectively, concurrent partnerships at year of migration, one year after migration, 2 years after migration, 3 years after migration, etc... until 20 years after migration or year of data collection, whichever came first, assessed up to 20 years. (data were collected with a life-event grid).
Evolution in occasional sexual partnerships after migration in France | At arrival in France, and then each year up to 20 years after arrival in France
  Proportion of the respondents who declared, retrospectively, occasional partnerships at year of migration, one year after migration, 2 years after migration, 3 years after migration, etc... until 20 years after migration or year of data collection, whichever came first, assessed up to 20 years. (data were collected with a life-event grid).
Evolution in transactional sexual partnerships after migration in France | At arrival in France, and then each year up to 20 years after arrival in France
  Proportion of the respondents who declared, retrospectively, transactional partnerships at year of migration, one year after migration, 2 years after migration, 3 years after migration, etc... until 20 years after migration or year of data collection, whichever came first, assessed up to 20 years. (data were collected with a life-event grid).

CONTACTS AND LOCATIONS:
Overall Officials: Annabel Desgrées du Loû, PhD, Principal Investigator — Institute of Research for Development, France

REFERENCES:
- [Derived] Vignier N, Dray Spira R, Pannetier J, Ravalihasy A, Gosselin A, Lert F, Lydie N, Bouchaud O, Desgrees Du Lou A, Chauvin P; PARCOURS Study Group. Refusal to provide healthcare to sub-Saharan migrants in France: a comparison according to their HIV and HBV status. Eur J Public Health. 2018 Oct 1;28(5):904-910. doi: 10.1093/eurpub/cky118. PMID 29982518
- [Derived] Gosselin A, Desgrees du Lou A, Lelievre E; PARCOURS Study Group. How to use sequence analysis for life course epidemiology? An example on HIV-positive Sub-Saharan migrants in France. J Epidemiol Community Health. 2018 Jun;72(6):507-512. doi: 10.1136/jech-2017-209739. Epub 2018 Feb 2. PMID 29437866
- [Derived] Pannetier J, Ravalihasy A, Lydie N, Lert F, Desgrees du Lou A; Parcours study group. Prevalence and circumstances of forced sex and post-migration HIV acquisition in sub-Saharan African migrant women in France: an analysis of the ANRS-PARCOURS retrospective population-based study. Lancet Public Health. 2018 Jan;3(1):e16-e23. doi: 10.1016/S2468-2667(17)30211-6. Epub 2017 Nov 23. PMID 29307383
- See also: web site of the Parcours study (in french) — http://www.parcours-sante-migration.com
- See also: Click here for more information about this study : the PARCOURS survey protocol (in english) — http://ceped.org/parcours/protocol-en.pdf